CLINICAL TRIAL: NCT05202834
Title: Evaluation of the UltraClear Laser Workstation for Skin Treatment - Histology Study of Laser Ablation on Human Skin
Status: Completed | Type: Observational
Sponsor: FA Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: UC 10-2021
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: UltraClear — Evaluation of the UltraClear Laser Workstation for Skin Treatment - Histology Study of Laser Ablation on human skin

SUMMARY:
Evaluation of the UltraClear Laser Workstation for Skin Treatment - Histology Study of Laser Ablation on human skin

DETAILED DESCRIPTION:
The study is being conducted to evaluate the safety and efficacy of the UltraClear Mid IR Fiber Laser Workstation using both superficial epidermis ablation capabilities and the deep ablative and coagulative capabilities into the dermis. Epidermis is the skin most outer layer that is supported by the dermis, which is the thick layer of living tissue below the epidermis which forms the true skin, containing blood capillaries, nerve endings, sweat glands, hair follicles, and other structures. Superficial ablative properties of the laser are the ability to remove thin and controlled layer of epidermis without damaging the underlaying layers of the skin, while the deep ablative properties of the laser are the ability to create a controlled and consistent mechanical and thermal injury in the skin that will lead to strong healing process that will improve the skin properties such as softness, elasticity and appearance. Round ø4.0 mm ( ~ø 1/8") Biopsies will be taken to examine the histologic effects of the treatments.

ELIGIBILITY:
Inclusion Criteria:

-1. Fitzpatrick skin type I-VI. 2. Male or female. 3. Subjects must be between 25 and 75 years of age. 4. Subjects must have ability to get treatment and biopsy from tissue in the abdomen or Buttock.

5. Subjects must read, understand, and sign the Informed Consent. 6. Subjects must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

1. Subjects must not have active localized or systemic infections.
2. Lidocaine or epinephrine allergy.
3. Subjects must not have a compromised ability for wound healing, such as: malnutrition, steroid use, history of collagen vascular disease (e.g. lupus, scleroderma, history of keloid scar formation), atrophic dermatitis or immunologic abnormalities such as vitiligo.
4. Subjects must not have had treatments with 5FU, hydroquinone, diclofenac, imiquimod, retinoids, or PDT within one month prior to enrollment.
5. Subjects must not currently be taking Accutane, or have taken Accutane within the last 6 months.
6. Subjects must not have a known allergy to the following topical products: lidocaine (numbing cream).
7. Subject must not have used topical steroids or retinoids within the last 3 months on treatment surfaces.
8. Subjects must not have a personal history of malignant melanoma, keloid scars, generalized psoriasis or systemic diseases that would preclude the use of topical anesthesia.
9. Subjects must agree to refrain from using cosmeceutical agents or topical agents during the course of the study, except as directed by study investigators.
10. Subjects must not be pregnant or breastfeeding.
11. Active sunburn or excessively tanned skin

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal and healthy Subjects
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Histology Study of Laser Ablation on human skin | Immediate after treatment
  Histological specimens microscope ready slides

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Assa, Study Director — FA Corporation
Locations (1):
- FA Corporation, Lincoln, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data